CLINICAL TRIAL: NCT05534451
Title: Comparison Among Three Different Video Scope Guided Nasotracheal Intubation: a Prospective, Non-randomised Controlled Trial
Brief Title: Comparison Among Three Different Video Scope Guided Nasotracheal Intubation.
Acronym: NTI
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other)
Responsible Party: Principal Investigator, Zhilin Wu, Principal Investigator, Union Hospital, Tongji Medical College, Huazhong University of Science and Technology
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2022SY
Record Dates: First submitted 2022-08-30; First posted 2022-09-09 (Actual); Last update posted 2023-08-18 (Actual); Status verified 2023-08

CONDITIONS: Intubation, Intratracheal; Airway Management
Keywords: nasotracheal intubation

STUDY DESIGN:
Intervention Model Description: According to the kinds of video methods uesd to assist in nasotracheal intubation, patients will be randomly divided into video laryngoscope group, video fiberoptic scope group and video rigid laryngoscope group, 20 participants in each group.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- video rigid laryngoscope group (Experimental): Similarly during intubation, the patient should be placed in the supine position with the neutral head. The endoscopic body of video rigid laryngoscope covered by a lubricated endotracheal tube enters the airway through the nasal cavity, then proceeds under visual conditions. When the epiglottis is exposed, if necessary, gently lift the patient's lower jaw so that the glottis is fully visible. The tube is pushed to approach and pass the glottis. Withdraw the endoscopic body while adjusting the depth of tube in the trachea. The intubation ends with tube fixation.
  Interventions: Behavioral: video rigid laryngoscope guided nasotracheal intubation
- video laryngoscope group (Experimental): First of all, participants will be asked to take supine position with neutral head. The operator will insert a lubricated endotracheal tube through the nasal cavity into the oropharynx, while he/she holds the handle of video laryngoscope in his/her left hand. Laryngoscope blade can be placed into oral cavity along the right corner of the patient's mouth, and the tongue is pushed to the left by moving the handle. Blade should arrive at a suitable depth to fully expose the epiglottis and glottis. After that, the operator can push the catheter with the right hand to approach and pass the glottis, sometimes Magill forceps are necessary. Finally, the tube is inserted into the trachea to the appropriate depth and fixed firmly.
  Interventions: Behavioral: video laryngoscope guided nasotracheal intubation
- video fiberoptic scope group (Experimental): It is suggested to apply paraffin oil to the surface of the insertion tube of video fiberoptic scope, where the friction with the inner wall of the endotracheal catheter will be reduced. The insertion tube together with a lubricated endotracheal tube will be placed into the nasopharynx through the nasal cavity of patient who takes supine position with neutral head. Push the insertion tube slowly and continuously along the airway until cuff passes through the glottis. Next carefully, the endotracheal tube can be delivered into the trachea, and the insertion tube can be withdrawn from the trachea. At last, the tracheal catheter can be fixed after the depth is adjusted to an appropriate level.
  Interventions: Behavioral: video fiberoptic scope guided nasotracheal intubation

INTERVENTIONS:
Behavioral: video laryngoscope guided nasotracheal intubation — According to the kinds of video methods uesd to assist in nasotracheal intubation, participants will be divided into video laryngoscope group. The data of the duration of catheter reaching oropharynx (T1), the duration of catheter reaching glottis (T2), successful intubation time (T3), the first-attempt intubation success rate, the total number of intubations for each participant, whether there is oral and nasal mucosa bleeding, whether the tracheal ring is pressed, whether the catheter is rotated, the heraodynamic changes, and the occurrence of throat complications within 2 hours after surgery, will be recorded respectively.
  Arms: video laryngoscope group
Behavioral: video rigid laryngoscope guided nasotracheal intubation — According to the kinds of video methods uesd to assist in nasotracheal intubation, participants will be divided into video rigid laryngoscope group. The data of the duration of catheter reaching oropharynx (T1), the duration of catheter reaching glottis (T2), successful intubation time (T3), the first-attempt intubation success rate, the total number of intubations for each participant, whether there is oral and nasal mucosa bleeding, whether the tracheal ring is pressed, whether the catheter is rotated, the heraodynamic changes, and the occurrence of throat complications within 2 hours after surgery, will be recorded respectively.
  Arms: video rigid laryngoscope group
Behavioral: video fiberoptic scope guided nasotracheal intubation — According to the kinds of video methods uesd to assist in nasotracheal intubation, participants will be randomly divided into video fiberoptic scope group. The data of the duration of catheter reaching oropharynx (T1), the duration of catheter reaching glottis (T2), successful intubation time (T3), the first-attempt intubation success rate, the total number of intubations for each participant, whether there is oral and nasal mucosa bleeding, whether the tracheal ring is pressed, whether the catheter is rotated, the heraodynamic changes, and the occurrence of throat complications within 2 hours after surgery, will be recorded respectively.
  Arms: video fiberoptic scope group

SUMMARY:
Nasotracheal intubation (NTI) has become the most optimal alternative to oral endotracheal intubation for oro-maxillofacial surgery because it can offer an excellent vision field of the mouth. Additional benefits include milder oropharynx stimulation, less airway secretions, and better tolerance for long term endotracheal intubation maintenance. Traditional NTI is performed under the guidance of indirect laryngoscope, which is often accompanied by longer maneuver time and adverse complications such as trauma and bleeding. The development of various visualization tools such as video laryngoscope, video fiberoptic scope and video rigid laryngoscope has greatly improved NTI. However, there is no consensus on which one is the best adjunctive device for NTI. Therefore, a study on a comparison of the clinical efficacy of the above three video scope guided methods for NTI will be conducted.

DETAILED DESCRIPTION:
A total of 60 eligible patients will be enrolled in this prospective study, they are scheduled to undergo elective oro-maxillofacial surgeries under general anaesthesia with nasotracheal intubation in the Union Hospital, Tongji Medical College, Huazhong University of Science and Technology. According to the kinds of video methods uesd to assist in nasotracheal intubation, patients will be randomly divided into video laryngoscope group, video fiberoptic scope group and video rigid laryngoscope group, 20 participants in each group. The data of the duration of catheter reaching oropharynx (T1), the duration of catheter reaching glottis (T2), successful intubation time (T3), the first-attempt intubation success rate, the total number of intubations for each participant, whether there is oral and nasal mucosa bleeding, whether the tracheal ring is pressed, whether the catheter is rotated, the heraodynamic changes, and the occurrence of throat complications within 2 hours after surgery, will be recorded respectively.

ELIGIBILITY:
Inclusion Criteria:

1. Participants scheduled for elective oro-maxillofacial surgery under general anesthesia.
2. Age between 18 and 65 years old.
3. The American Society of Anesthesiologists (ASA) Ⅰ～Ⅱ.
4. Body mass index (BMI) 18.5～24.9kg/m2.
5. Mallampati Ⅰ～Ⅱ.
6. Able to give informed consent.

Exclusion Criteria:

1. Participants with severe intranasal diseases.
2. Participants with severe and uncontrolled clotting diseases.
3. Participants with skull base fractures and cerebrospinal fluid leakage.
4. Participants with unstable cardiovascular and cerebrovascular diseases, or with poor tolerance to vagal stimulation.
5. Participants who are deemed ineligible for participation in the clinical trial by the investigator.
6. Participants who have to receive the alternative therapy to establish ventilation after the several attempts for nasotracheal intubation.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-09-01 (Estimated); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-07-31 (Estimated)

PRIMARY OUTCOMES:
the duration of catheter reaching oropharynx | within 1 minute
  time requirements for delivering the anterior segment of the endotracheal tube from the nasal cavity to the oropharynx
the duration of catheter reaching glottis | within 1 minute
  time requirements for the anterior segment of the endotracheal tube from being put into the nasal cavity to the glottis being exposed
successful intubation time | within 3 minute
  time requirements for delivering the anterior segment of the endotracheal tube from the nasal cavity to the trachea
the first-attempt intubation success rate | anticipated eight months
  number of successful first-attempt intubation/total number of intubations
average number of intubations | anticipated eight months
  average number of nasotracheal intubations for each participant

SECONDARY OUTCOMES:
the number of participants whose oral and nasal mucosa bleeds during intubation | within 3 minute
  during nasotracheal intubation, whether airway soft tissue is damaged, such as bleeding
the number of participants whose tracheal ring is pressed and catheter is rotated when intubation | within 3 minute
  during nasotracheal intubation, record whether the operator presses the tracheal ring and rotates the tracheal tube to assist intubation
Blood pressure values before and after intubation intubation | 20 minute
  record blood pressure values before and after intubation
Heart rate values before and after intubation intubation | 20 minute
  record heart rate before and after intubation
the occurrence of throat complications | within 2 hours after surgery
  inquiry and record intubation related complications, such as sore throat and hoarseness

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Park DH, Lee CA, Jeong CY, Yang HS. Nasotracheal intubation for airway management during anesthesia. Anesth Pain Med (Seoul). 2021 Jul;16(3):232-247. doi: 10.17085/apm.21040. Epub 2021 Jul 30. PMID 34352965
- [Background] Zhang J, Lamb A, Hung O, Hung C, Hung D. Blind nasal intubation: teaching a dying art. Can J Anaesth. 2014 Nov;61(11):1055-6. doi: 10.1007/s12630-014-0223-9. Epub 2014 Aug 15. No abstract available. PMID 25125251
- [Background] Gorback MS. Inflation of the endotracheal tube cuff as an aid to blind nasal endotracheal intubation. Anesth Analg. 1987 Sep;66(9):916-7. No abstract available. PMID 3619105
- [Background] Abdallah R, Galway U, You J, Kurz A, Sessler DI, Doyle DJ. A randomized comparison between the Pentax AWS video laryngoscope and the Macintosh laryngoscope in morbidly obese patients. Anesth Analg. 2011 Nov;113(5):1082-7. doi: 10.1213/ANE.0b013e31822cf47d. Epub 2011 Sep 14. PMID 21918156
- [Background] Tachibana N, Niiyama Y, Yamakage M. Less postoperative sore throat after nasotracheal intubation using a fiberoptic bronchoscope than using a Macintosh laryngoscope: A double-blind, randomized, controlled study. J Clin Anesth. 2017 Jun;39:113-117. doi: 10.1016/j.jclinane.2016.10.026. Epub 2017 Apr 6. PMID 28494884
- [Background] Enterlein G, Byhahn C; American Society of Anesthesiologists Task Force. [Practice guidelines for management of the difficult airway: update by the American Society of Anesthesiologists task force]. Anaesthesist. 2013 Oct;62(10):832-5. doi: 10.1007/s00101-013-2222-6. German. PMID 24104949
- [Background] Park EY, Kim JY, Lee JS. Tracheal intubation using the Airtraq: a comparison with the lightwand. Anaesthesia. 2010 Jul;65(7):729-32. doi: 10.1111/j.1365-2044.2010.06376.x. Epub 2010 May 17. PMID 20497149